CLINICAL TRIAL: NCT00572364
Title: A Phase I, Open-label, Dose Escalation Study to Assess the Safety and Tolerability of AZD2281 Following Single and Multiple Oral Doses in Patients in Japan With Advanced Solid Malignancies
Brief Title: Open Label, Dose Escalation Phase I Study of AZD2281
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D0810C00001
Record Dates: First submitted 2007-12-12; First posted 2007-12-13 (Estimated); Last update posted 2009-08-20 (Estimated); Status verified 2009-08

CONDITIONS: Advanced Solid Malignancies
Keywords: Cancer; Advanced solid malignancies
MeSH Terms: conditions — Neoplasms | interventions — olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: KU-0059436 (AZD2281)(PARP inhibitor) — oral
  Other Names: Olaparib

SUMMARY:
The purpose of the study is to assess the safety and tolerability of AZD2281 following single and multiple oral doses in patients in Japan with advanced solid malignancies

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed malignant solid tumour and refractory to standard therapy or for which no suitable effective standard therapy exists.

Exclusion Criteria:

* Patients undergone, within 4 weeks prior to trial entry, an anti-cancer therapy which includes chemotherapy (or a longer period depending on the defined characteristics of the drugs used eg,. 6 weeks for mitomycin C or nitrosourea.

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2007-11; Primary Completion 2009-03 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to determine the safety and tolerability of AZD2281. | assessed after each visit

SECONDARY OUTCOMES:
The secondary objectives of the study are to determine MTD and pharmacokinetic profile of oral AZD2281. | assessed after each visit

CONTACTS AND LOCATIONS:
Overall Officials: James Carmichael, Study Director — KuDOS/AstraZeneca
Locations (1):
- Research Site, Tokyo, Japan

REFERENCES:
- [Derived] Yamamoto N, Nokihara H, Yamada Y, Goto Y, Tanioka M, Shibata T, Yamada K, Asahina H, Kawata T, Shi X, Tamura T. A Phase I, dose-finding and pharmacokinetic study of olaparib (AZD2281) in Japanese patients with advanced solid tumors. Cancer Sci. 2012 Mar;103(3):504-9. doi: 10.1111/j.1349-7006.2011.02179.x. Epub 2012 Jan 30. PMID 22145984